CLINICAL TRIAL: NCT02360735
Title: Manual Lymph Drainage for Patients With Acute Total Knee Replacement
Brief Title: Manual Lymph Drainage
Acronym: MLD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Anne Arundel Health System Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLD-2014
Record Dates: First submitted 2015-01-29; First posted 2015-02-11 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Total Knee Arthroplasty; Post-operative Edema
MeSH Terms: interventions — Manual Lymphatic Drainage; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients randomized to this arm will follow the current standard for post-operative care.
  Interventions: Other: Physical Therapy
- Experimental (Experimental): Patients randomized to this arm will follow the current standard for post-operative care as well as 2 daily sessions of manual lymphatic drainage.
  Interventions: Other: Manual Lymphatic Drainage; Other: Physical Therapy

INTERVENTIONS:
Other: Manual Lymphatic Drainage — Manual Lymphatic Drainage (MLD) is a specialized massage technique utilized to decrease various forms of edema. This technique promotes reuptake of interstitial fluid along the pathways of the lymphatic system. This technique promotes healing, decrease swelling, and decrease pain.
  Other Names: MLD; Manual Lymph Drainage
  Arms: Experimental
Other: Physical Therapy — All patients will participate in joint physical therapy classes during their inpatient stay.

SUMMARY:
Manual Lymphatic Drainage (MLD) is a specialized massage technique utilized to decrease various forms of edema. This technique promotes reuptake of interstitial fluid along the pathways of the lymphatic system. This technique promotes healing, decrease swelling, and decrease pain.

DETAILED DESCRIPTION:
Manual Lymphatic Drainage (MLD) is a specialized massage technique utilized to decrease various forms of edema. Edema can limit function, range of motion (ROM) and increase pain after surgery. Studies have shown that decreasing edema can increase knee strength and functional performance on various standardized measures. MLD has been shown to be effective in patients with hind foot operations and increases ROM post total knee replacement (TKR) surgery. The aim of this study is to determine whether MLD on a sample of patients with TKR will decrease edema, increase ROM and decrease pain as compared to TKR patients who do not receive MLD.

ELIGIBILITY:
Inclusion Criteria:

* s/p total knee replacement
* Primary diagnosis of osteoarthritis or degenerative joint disease
* Able to read and understand English to consent
* Acceptance of the study protocol procedure

Exclusion Criteria:

* Active infection
* Tumor
* Metastatic or systemic malignancy
* Acute thrombus
* History of pulmonary embolism
* Major cardiac pathology such has angina
* Heart attack or uncompensated congestive heart failure (CHF)
* Body mass index (BMI) > 40
* Pregnant or lactating women
* Renal dysfunction
* Joint revision
* Hospitalization length of stay less than or greater than 3 days
* Previous knee replacement
* Bilateral knee replacement

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 3 days
  Determine if performing MLD after TKR surgery decreases pain in the knee as compared to controls
Range of Motion | 3 days
  Determine if performing MLD after TKR surgery increases range of motion as compared to the standard of care
Girth | 3 days
  Determine if performing MLD after TKR surgery decreases girth and swelling in the knee as compared to the standar of care

CONTACTS AND LOCATIONS:
Overall Officials: Paul King, M.D., Principal Investigator — Anne Arundel Medical Center, OSMC
Locations (1):
- Anne Arundel Medical Center, Annapolis, Maryland, United States

REFERENCES:
- [Background] Kessler T, de Bruin E, Brunner F, Vienne P, Kissling R. Effect of manual lymph drainage after hindfoot operations. Physiother Res Int. 2003;8(2):101-10. doi: 10.1002/pri.277. PMID 12879732
- [Background] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725
- [Background] Ebert JR, Joss B, Jardine B, Wood DJ. Randomized trial investigating the efficacy of manual lymphatic drainage to improve early outcome after total knee arthroplasty. Arch Phys Med Rehabil. 2013 Nov;94(11):2103-11. doi: 10.1016/j.apmr.2013.06.009. Epub 2013 Jun 26. PMID 23810354
- [Background] Shimoyama Y, Sawai T, Tatsumi S, Nakahira J, Oka M, Nakajima M, Jotoku T, Minami T. Perioperative risk factors for deep vein thrombosis after total hip arthroplasty or total knee arthroplasty. J Clin Anesth. 2012 Nov;24(7):531-6. doi: 10.1016/j.jclinane.2012.02.008. Epub 2012 Sep 21. PMID 23006595
- [Background] Watanabe H, Sekiya H, Kariya Y, Hoshino Y, Sugimoto H, Hayasaka S. The incidence of venous thromboembolism before and after total knee arthroplasty using 16-row multidetector computed tomography. J Arthroplasty. 2011 Dec;26(8):1488-93. doi: 10.1016/j.arth.2011.01.001. Epub 2011 Feb 12. PMID 21316910
- [Background] Januel JM, Chen G, Ruffieux C, Quan H, Douketis JD, Crowther MA, Colin C, Ghali WA, Burnand B; IMECCHI Group. Symptomatic in-hospital deep vein thrombosis and pulmonary embolism following hip and knee arthroplasty among patients receiving recommended prophylaxis: a systematic review. JAMA. 2012 Jan 18;307(3):294-303. doi: 10.1001/jama.2011.2029. PMID 22253396